CLINICAL TRIAL: NCT04373499
Title: A Randomized Clinical Trial Evaluating the Effectiveness of Virtual Teach-to-Goal Education vs. Brief Intervention for Children
Brief Title: Virtual Teach-to-Goal Education vs. Brief Education for Children
Acronym: V-TTG vs BI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: American College of Chest Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-1080
Record Dates: First submitted 2018-11-09; First posted 2020-05-04 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Asthma; Bronchospasm; Shortness of Breath
Keywords: Inhaler; Education; Asthma; Learning; Module; Virtual Teach to Goal
MeSH Terms: conditions — Asthma; Bronchial Spasm; Dyspnea | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: We will conduct a single-site randomized clinical trial of V-TTG versus brief intervention (BI) for school-aged children (5-11 years) with severe asthma hospitalized at University of Chicago Comer Children's Hospital. We aim to enroll 70 participants. The project team will identify eligible children who meet inclusion criteria. Block randomization will be utilized, stratified by age (5-8 vs. 9-11 years).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Teach-to-Goal (V-TTG) (Experimental): The RA will show the patient how to use the tablet to access the education module and be available for questions about the technology / tablet but not about the content. Within the module, the child will:
  * answer questions about how to use the inhaler as part of a pre-video assessment.
  * watch a video about how to correctly use a Metered Dose Inhaler (MDI) and spacer.
  * answer questions on the tablet to assess how well they understand how to use the inhaler.
  If a child answers any questions incorrectly, they will watch the video again and have another chance to answer the incorrect questions. The child will receive instruction by video one or multiple times (up to 3 times), depending on how much they understand after each round of instruction, as demonstrated by their responses to questions.
  Interventions: Behavioral: Virtual Teach to Goal
- Brief Intervention (BI) (Active Comparator): The RA will give the patient a handout about inhaler technique and read the steps to the child.
  Interventions: Behavioral: Brief Intervention

INTERVENTIONS:
Behavioral: Virtual Teach to Goal — Virtual Teach-to-Goal is an educational module that teaches children how to use their inhaler properly; this is done with an IPAD. In the module, the child will complete a series of questions as a pre-assessment, watch a video about how to use the inhaler properly, and then answer a series of questions as a post-assessment. If a child answers any questions incorrectly, they will watch the video again and have another chance to answer the incorrect questions. The child will receive instruction by video one or multiple times (up to 3 times), depending on how much they understand after each round of instruction, as demonstrated by their responses to questions.
  Other Names: VTTG
  Arms: Virtual Teach-to-Goal (V-TTG)
Behavioral: Brief Intervention — There is a handout that describes proper inhaler technique. The RA reads the handout to the child.
  Other Names: BI
  Arms: Brief Intervention (BI)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of two different ways to teach hospitalized children how to use a metered dose inhaler and to follow-up after discharge home from the hospital to determine durability of the education.

DETAILED DESCRIPTION:
Asthma is the most common chronic childhood condition and has significant adverse consequences. One in 12 United States children has asthma, resulting in 13.4 million missed school days, 1 million emergency department visits, and 140,000 hospitalizations annually.

A key barrier to self-management of asthma is improper use of respiratory inhalers, which limits disease control. Better inhaler technique is associated with improved asthma outcomes for children. Assessment and education of inhaler technique are recommended at all healthcare encounters, however it is limited in practice because it is resource intensive (both personnel and time) and lacks fidelity. Thus, low-resource interventions that accurately teach inhaler skills are needed to impact pediatric asthma outcomes.

Teach-to-Goal (TTG) is a patient-centered strategy that uses tailored rounds of teaching and assessments to ensure mastery of inhaler technique. Studies show it is effective but resource intensive. A "virtual TTG" (V-TTG) intervention represents an opportunity to deliver inhaler technique education with a high-fidelity, low-resource, and feasible strategy. The module utilizes innovative learning technology with video demonstrations and assessment questions to tailor education to each user; the cycles of assessment and education continues until satisfactory mastery is achieved.

This study evaluates the comparative effectiveness of this high-fidelity, low-resource, and feasible model (V-TTG) versus a standardized brief intervention that mimics usual care to deliver tailored inhaler technique education to children with severe asthma via a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. The child is between the ages of 5-10 years old
2. The child is admitted for an asthma exacerbation, wheezing, or bronchospasm
3. The child is admitted to the Pediatric Hospital Medicine Service at Comer Children's Hospital
4. The child is prescribed albuterol

Exclusion Criteria:

1. The child/parent decline or unable to provide consent/assent, do not speak/read English
2. The child cannot use an inhaler by themselves without a mask
3. The child previously participated in this study
4. The child is currently in the pediatric intensive care unit (PICU)

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with metered dose inhaler (MDI) misuse immediately after V-TTG vs. BI education | Initial study visit / baseline
  Evaluate effectiveness of V-TTG as compared to BI as measured by inhaler technique post-intervention. This will provide data on the short-term effectiveness of the interventions. Each patient's inhaler technique will be assessed using validated inhaler checklists by the trained assessor.

SECONDARY OUTCOMES:
Acceptability of V-TTG among children and parents based on Likert-scale questions (1-5) | Initial study visit - after completing V-TTG intervention
  Questionnaires of children and parents immediately after completing the V-TTG intervention. Likert-scale questions will focus on whether children and parents like the V-TTG education, would be willing to use, and would recommend to a friend.
Usability of V-TTG among children and parents based on open-ended questions | Initial study visit - after completing V-TTG intervention
  Interviews with children and parents immediately after completing the V-TTG intervention. Open-ended questions will be utilized to assess what children and parents like or do not like about the module and how it could be utilized in clinical settings, at home, at school.
Proportion of participants with metered dose inhaler (MDI) misuse in VTTG vs BI arms at 1 month after education | Follow-up visit at 1 month
  Retention of proper inhaler technique skills
Self-efficacy: Questionnaire | Initial study visit - at baseline and immediately after intervention
  Questionnaire with Likert-scale questions (1-5) to assess self-efficacy about inhaler technique pre vs post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Volerman A, Balachandran U, Zhu M, Akel M, Hull A, Siros M, Luna V, Xu I, Press VG. Evaluating inhaler education interventions for hospitalized children with asthma: A randomized controlled trial. Ann Allergy Asthma Immunol. 2023 Aug;131(2):217-223.e1. doi: 10.1016/j.anai.2023.02.023. Epub 2023 Mar 3. PMID 36870528